CLINICAL TRIAL: NCT03337282
Title: Incidence and Characteristics of Postoperative Cognitive Dysfunction in Elderly Quebec Francophone Patients Following Major Surgery Under Standardized General Anesthesia With Tight Hemodynamic Control: A Prospective Observational Study
Brief Title: Incidence and Characteristics of Postoperative Cognitive Dysfunction in Elderly Quebec Francophone Patients
Status: Terminated | Type: Observational
Why Stopped: Elderly population difficult to recruit
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Professor, DIrector of Research, Department of Anesthesiology, Université de Montréal, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2018-1197
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Delirium; Cognitive Impairment; Cognitive Decline; Cognitive Change; Postoperative Cognitive Dysfunction; Postoperative Delirium
Keywords: anesthesia; noncardiac surgery; major surgery; POCD
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: Adults 70 years of age or older undergoing major noncardiac surgery under protocolized general anesthesia
  Interventions: Procedure: Protocolized general anesthesia

INTERVENTIONS:
Procedure: Protocolized general anesthesia — Induction and maintenance of general anesthesia, post-operative analgesia with protocolized drugs and doses. Maintenance of MAP +/- 20% of baseline with vasopressors as needed.

SUMMARY:
The purpose of this study is to determine what percentage of patients have cognitive problems (for example, memory or concentration difficulties) after surgery and anesthesia, what the characteristics of these problems are, and whether they persist over time. In particular, the investigators want to study this in the French-speaking Quebec population with cognitive evaluation tools adapted for this population.

DETAILED DESCRIPTION:
Multiple experimental and observational studies have established that a non-negligible percentage of individuals undergoing surgery and anesthesia will experience a postoperative decline in mental abilities. These cognitive changes can range from postoperative delirium to more subtle and longer lasting (weeks to months) impairments; these latter changes are often referred to in the literature as postoperative cognitive dysfunction (POCD). While the precise causes of POCD remain nebulous, a clear epidemiological risk factor is advanced age - a demographic group that accounts for an increasing percentage of elective surgeries in North America. Several RCTs have attempted to link specific aspects of anesthesia, such as depth of anesthesia, regional vs general anesthesia, hemodynamic parameters, specific anesthetic agents, etc., to the risk of developing POCD in both the elderly and general populations. Results have often been conflicting and, based on current evidence, it is difficult to identify any specific anesthetic strategy that clearly reduces the risk of POCD. The present study aims to establish the incidence and neuropsychological characteristics of POCD in the investigator's local patient population as well as to establish the feasibility of pre- and postoperative cognitive testing with assessment tools adapted to and validated for Quebec francophones in order to lay the groundwork for future studies by the research group of interventions targeting specific anesthetic techniques and monitoring modalities.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* Undergoing elective abdominal, gynecological, or urological surgery requiring post-operative hospitalization and with an expected anesthesia time of 60 minutes or more
* Seen in pre-operative clinic of Maisonneuve-Rosemont hospital

Exclusion Criteria:

* Known dementia or other cognitive impairment
* Psychiatric disease
* Significant hearing or vision impairment
* Inability to communicate in French
* Allergy or other contraindication to medications in standardized anesthesia protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly Quebec francophone patients undergoing elective major non-cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Post-operative cognitive dysfunction | Baseline cognitive testing will be performed before surgery, then repeated on day before discharge or post-operative day 7 and then again at approximately post-operative day 30.
  Presence of post-operative cognitive dysfunction as determined by neuropsychological tests. A diagnosis of POCD will be made under the follow circumstances: a) A decrease in score from one assessment to the next (e.g., postoperatively vs. preoperatively) that results in the subject changing from within normal limits to below normal limits on the Montreal Cognitive Assessment (MoCA) b) A decrease in score of ≥ 1 standard deviation on the normed tests (MoCA, verbal fluency

SECONDARY OUTCOMES:
Post-operative delirium | Post-operative days 1 and 2
  Participants will be assessed for delirium via administration of the Confusion Assessment Method
Self-assessment of applied cognitive abilities | Pre-operatively, then post-operatively on day before discharge or post-operative day 7, then again on approximately post-operative day 30
  The PROMIS self-assessment questionnaire "Applied cognition - Abilities" will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebé, MD, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saffer BY, Lanting SC, Koehle MS, Klonsky ED, Iverson GL. Assessing cognitive impairment using PROMIS((R)) applied cognition-abilities scales in a medical outpatient sample. Psychiatry Res. 2015 Mar 30;226(1):169-72. doi: 10.1016/j.psychres.2014.12.043. Epub 2015 Jan 8. PMID 25639374
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Inouye SK, Kosar CM, Tommet D, Schmitt EM, Puelle MR, Saczynski JS, Marcantonio ER, Jones RN. The CAM-S: development and validation of a new scoring system for delirium severity in 2 cohorts. Ann Intern Med. 2014 Apr 15;160(8):526-533. doi: 10.7326/M13-1927. PMID 24733193
- [Background] St-Hilaire A, Hudon C, Vallet GT, Bherer L, Lussier M, Gagnon JF, Simard M, Gosselin N, Escudier F, Rouleau I, Macoir J. Normative data for phonemic and semantic verbal fluency test in the adult French-Quebec population and validation study in Alzheimer's disease and depression. Clin Neuropsychol. 2016 Oct;30(7):1126-50. doi: 10.1080/13854046.2016.1195014. Epub 2016 Jun 9. PMID 27279436
- [Background] Howland M, Tatsuoka C, Smyth KA, Sajatovic M. Evaluating PROMIS((R)) applied cognition items in a sample of older adults at risk for cognitive decline. Psychiatry Res. 2017 Jan;247:39-42. doi: 10.1016/j.psychres.2016.10.072. Epub 2016 Nov 1. PMID 27863317
- [Background] Vercambre MN, Cuvelier H, Gayon YA, Hardy-Leger I, Berr C, Trivalle C, Boutron-Ruault MC, Clavel-Chapelon F. Validation study of a French version of the modified telephone interview for cognitive status (F-TICS-m) in elderly women. Int J Geriatr Psychiatry. 2010 Nov;25(11):1142-9. doi: 10.1002/gps.2447. PMID 20054838